CLINICAL TRIAL: NCT05248828
Title: Testing of New Method in Sanitizing Breast Pump Equipment in the NICU
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: IRB1750118
Record Dates: First submitted 2022-01-26; First posted 2022-02-21 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Breast Pumping
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate a newly developed device, Q. Basin. The Q. Basin is a multifunctional, single patient use device that can sanitize breast pump parts, bottles, and reusable feeding devices for patients admitted under one year of age. Improving the current sanitation method would provide a quick and efficient sanitation process for breast pump parts. This study will compare the Q. Basin to the current method of steam bag sanitation.

DETAILED DESCRIPTION:
Firstly, 10 participant's breast pump parts are collected, divided, washed, and dried before comparing the two methods of steam sanitation. We will test to compare the safety of the Q. Basin compared to the current method of steam bag sanitation. We will collect participant's breast pump parts and complete surface swab testing for bacteria and mold immediately after sanitation and additionally 24 hours later.

Secondly, 20 participant questionnaires will measure satisfaction ratings of participants pumping human milk for hospitalized infants using two different wash, dry and steam sanitation methods. This study design will determine if participant satisfaction improves with breast pump part sanitation using the Q. Basin, compared to the current steam sanitization bag method.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who are pumping human milk for hospitalized infants in the Neonatal Intensive Care Unit.

Exclusion Criteria:

* Mothers under the age of 18 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers who are pumping human milk for hospitalized infants in the Neonatal Intensive Care Unit
Study Population: In the Neonatal Intensive Care Unit, mothers who wish to pump human milk for their hospitalized infant do so with an electric breast pump. All 10 breast pump parts are used to pump human milk 8-10 times a day. After each pumping session, breast pump parts that contact human milk are washed and air-dried thoroughly until next use. Once a day, clean pump parts are placed in a sanitation bag and steam sanitized in the microwave.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Safety Rate | Immediately after steam bag sanitation
  The Safety rate between the Q. Basin and steam bag sanitation is measured by surface swab testing
Safety Rate | 24 hours later
  The Safety rate between the Q. Basin and steam bag sanitation is measured by surface swab testing

SECONDARY OUTCOMES:
Satisfaction Rate Questionnaire | At the end of 2 cycles (each cycle is 3 hours) of steam bag sanitation
  The satisfaction rate is measured by participants comparing two different methods of breast pump part sanitation

CONTACTS AND LOCATIONS:
Overall Officials: Marron, Principal Investigator — Nemours Childrens Health- Delaware
Locations (1):
- Nemours Childrens Hospital Delaware, Wilmington, Delaware, United States